CLINICAL TRIAL: NCT02656563
Title: Phase II, Randomized, Open Label to Evaluate Efficacy,Safety of Radium 223 in Prolonging the Off Treatment Interval in Men With Rising PSA Post-rad, or Post-prostatectomy Without Bone Mets on Intermittent Androgen Ablation Therapy
Brief Title: Radium 223 Following Intermittent ADT
Acronym: RAND
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Urology Research Consortium (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CURC-004; 17848 (Other: Bayer)
Record Dates: First submitted 2015-11-05; First posted 2016-01-15 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radium 223 Arm (Experimental): Radium 223 Dichloride (Xofigo®)
  Interventions: Radiation: Radium 223 Dichloride (Xofigo®)
- Non Treatment Arm (No Intervention): Control Arm

INTERVENTIONS:
Radiation: Radium 223 Dichloride (Xofigo®) — Radium 223 Dichloride (Xofigo®) monthly for six months
  Other Names: Xofigo®
  Arms: Radium 223 Arm

SUMMARY:
This is a multicentre, phase II, randomized, open label study to evaluate the efficacy and safety of monthly Radium 223 in prolonging the off treatment interval of men with localized prostate cancer receiving intermittent androgen ablation therapy for a rising PSA post-radiation or post-prostatectomy, who are at high risk for occult metastases.

DETAILED DESCRIPTION:
Eligible subjects will be randomized in a 1:1 ratio to receive either (1) study medication, Radium 223 monthly for six months or (2) no treatment (usual care). All patients will have a physical exam, PSA, testosterone and clinical lab tests conducted monthly. Group 1 will receive monthly Radium 233 beginning one month after discontinuing ADT, for a maximum of 6 months of treatment. Radium-223 will be given in accordance with the Canadian product label and Product Monograph at 50kBq/kg.

If PSA reaches 5ng/ml before 7 months after discontinuing ADT, the patient will discontinue Radium 223 and resume ADT. Group 2 will have no further therapy until their PSA reaches 5ng/ml, at which point they will resume ADT.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and write (health outcome questionnaires are self- administered), understand instructions related to study procedures and to give written informed consent.
2. Age ≥ 45 and ≤ 85 years.
3. Histologically documented diagnosis (including Gleason grade) of adenocarcinoma of the prostate.
4. Subject has received external beam radiation, brachytherapy or radical prostatectomy for the treatment of localized prostate cancer, or is being treated with primary androgen deprivation.
5. Subject has completed intermittent androgen ablation therapy or is about to complete ADT.
6. Patients treated with brachytherapy must be at least 3 years post implant.
7. Subject meets both of the following criteria:

   * PSA >5.0 and < 100 ng/ml and rising on 2 successive occasions at least one month apart prior to ADT. PSA must be < 2.0 after 6-8 months of ADT (+/- 4 weeks). At month 8 (or within 4 weeks after month 8), following documentation that PSA <2.0, patients will be entered.
   * Patients must also have two of the following high risk criteria:

     * Primary Gleason score >8
     * Baseline PSA > 20 ng/ml (pre-treatment)
     * PSA recurrence > 0.2 within 1 year (post RP)
     * PSA DT prior to ADT < 6 months
     * PSA > 1.0 ng/ml after 8 months of ADT
8. Adequate hematological, liver, and renal function including:

   * Absolute neutrophil count (ANC) ≥ 1.5 x109/L
   * Platelet count ≥ 100 x109/L
   * Hemoglobin ≥10.0 g/dL (100 g/L; 6.2 mmol/L)
   * Total bilirubin level ≤ 1.5 x institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
   * Albumin > 25 g/L
9. Eastern Cooperative Oncology Group Performance (ECOG) performance 0 or 1 (Appendix 2).
10. Negative bone scan and negative CT scan for visceral (extra nodal) mets within 12 months of study entry. Bone scan and CT may be performed after initiation of ADT. If lymphadenopathy present, must be <3 cm in shortest diameter.
11. Able to swallow and retain oral medication.
12. Able and willing to participate in the full study.
13. Willingness to use condoms if sexually active.

Exclusion Criteria:

1. Previous treatment for prostate cancer with any of the following:

   * Chemotherapy
   * Hormonal therapy (e.g. megestrol, medroxyprogesterone, cyproterone, DES) within the previous year. (Note: Patients who are on their first cycle of intermittent androgen deprivation therapy within 8 months of initiating treatment are eligible).
   * Glucocorticoids (except inhaled or topical) within the previous 3 months.
   * Ketoconazole
2. Concurrent and previous use within 3 months of the following medications:

   * Finasteride
   * Dutasteride
   * Any investigational 5α-reductase inhibitors
   * Anabolic steroids
   * Medications with anti-androgenic properties such as cimetidine.
3. Patients may not be receiving any other investigational agents within 30 days prior to the first dose of study drug or anytime during the study period.
4. Subject currently has evidence of distant metastases on bone scan, or visceral metastases on CT scan. Patients with bulky LN mets. (> 3 cm in shortest diameter). (Note: Adenopathy < 3 cm in shortest diameter is not an exclusion criterion).
5. Subject has received adjuvant or neoadjuvant androgen ablation within the previous 12 months.
6. Any unstable serious co-existing medical condition(s) including but not limited to uncontrolled diabetes, peptic ulcer disease, Crohn's disease and ulcerative colitis.
7. Abnormal liver function tests (alkaline phosphatase [ALP], alanine aminotransferase [ALT], aspartate aminotransferase [AST]) > 2.5 times upper limit of normal (ULN) or bilirubin > 1.5 times ULN)
8. Previous malignancy (not including curatively treated basal or squamous cell carcinoma of the skin within the previous 2 years or Ta bladder cancer with negative surveillance cystoscopy within the past year).
9. History or current evidence of drug or alcohol abuse within the past 12 months.
10. History of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the subject. This includes:

    * Imminent spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI). Patients with history of spinal cord compression should have completely recovered.
    * Any infection ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 Grade 2
    * Cardiac Failure New York Heart Association (NYHA) Class III or IV
    * Bone marrow dysplasia
    * Fecal incontinence
11. Prior hemibody external radiotherapy, or systemic therapy with radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188, or radium-223 dichloride).

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
PSA > 5.0ng/ml | Time to PSA > 5.0ng/ml in the off treatment, through study completion at 2 years.
  Time to PSA > 5.0ng/ml in the off treatment interval during intermittent androgen ablation therapy, as measured from randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Klotz, MD, Study Chair — Canadian Urology Research Consortium
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada